CLINICAL TRIAL: NCT03684707
Title: Cancer Chemoprevention by Metformin Hydrochloride Compared to Placebo in Oral Potentially Malignant Lesions: A Randomised Clinical Trial
Brief Title: Cancer Chemoprevention by Metformin Hydrochloride Compared to Placebo in Oral Potentially Malignant Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Nasr, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cairo University
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Metformin; Starch

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin Hcl 500Mg 24Hr Sa Tab (Active Comparator): Metformin Hcl 500Mg 24Hr Sa Tab drug is given to the patient
  Interventions: Drug: Metformin Hcl 500Mg 24Hr Sa Tab
- control (Placebo Comparator): starch tablets
  Interventions: Other: starch tablet

INTERVENTIONS:
Drug: Metformin Hcl 500Mg 24Hr Sa Tab — Glucophage 500 mg once daily
  Other Names: Glucophage
  Arms: Metformin Hcl 500Mg 24Hr Sa Tab
Other: starch tablet — starch tablets
  Arms: control

SUMMARY:
Evaluation of the metformin drug effect as a drug that found to improve the quality of tissues, decrease signs & symptoms of cancer, and decrease histo-pathological criteria of dysplasia.

This will be done by the aid of measuring salivary Micro RNA 31 & 210 in saliva in addition to measure cyclin A2 as an immuno-histochemical analysis.

DETAILED DESCRIPTION:
Oral squamous cell carcinomas (OSCCs) are among the most common types of head and neck cancers and are a major cause of significant morbidity. It was reported that 16- 62% of OSCCs develop from premalignant lesions, which often presents clinically as white or red mucosal patches known as leukoplakia and erythroplakia. The role of miRNA in cancer has been reiterated and established by many studies that have shown that miRNA signatures (i.e., mRNA expression profiles) can be useful for classifying human cancers. These studies have identified "cancer related miRNAs" through investigating expression profiles in matched normal and tumor tissues, as well as in body fluids. In addition, a vast number of studies have shown that miRNAs can play a role in regulating the expression of oncogenes and tumor suppressor genes, whereas others have shown that miRNA gene deletion or mutation can lead cancer initiation, progression and metastasis . Several potential mechanisms have been suggested for the ability of metformin to suppress cancer growth in vitro and vivo:

(1) Activation of LKB1/AMPK pathway, (2) Induction of cell cycle arrest and/or apoptosis, (3) Inhibition of protein synthesis, (4) Reduction in circulating insulin levels, (5) Inhibition of the unfolded protein response (UPR), (6) Activation of the immune system.

This study is performed to evaluate metformin effect on the patients premalignant lesion versus maintenace follow ups.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age range from 20 to 70 years.
* Patients able to return for the follow up visits and can perform oral hygiene measures.
* Clinically diagnosed and histologically confirmed as having oral potentially malignant lesions.
* Patients agreed to sign a written consent after understanding the nature of the study
* Patients have diagnosed oral premalignant lesion/lesions and not yet turned into malignancy (atrophic lichen planus- leukoplakia-erythroplakia - oral submucous fibrosis)

Exclusion Criteria:

* - Diabetic patients (Diabetes Mellitus Type I & II)
* Patients have cardiovascular, lung, Renal, Liver diseases
* Patients on H2 blocker & proton pump inhibitors therapy as Ranitidine (affects metformin absorption and clearance)
* Those with allergy or sensitivity to Metformin or Retinoids therapy or having any contraindication for their use.
* Systemic and/or local systemic drug therapy within the last 3 months prior to the start of the study
* Patients on steroidal or Non-steroidal anti-inflammatory drugs (NSAIDs) for at least the last 6 months
* Patients on Antibiotics treatment for at least the last 2 months
* Patients on Retinoid, green tea supplements or another natural products therapy
* Patients with already diagnosed malignant lesion/lesions
* Pregnant or Lactating females
* Vulnerable groups as prisoners, mentally disabled, etc…

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate lesion size in millimeters | 1 year
  Evaluate lesion size in millimeters

SECONDARY OUTCOMES:
Measurement of salivary Micro RNA | 1 year
  measuring salivary markers 31& 210 in saliva and also in tissue biopsy
Measuring immuno-histochemical marker | 1 year
  Measuring cyclin A2 marker in tissues

CONTACTS AND LOCATIONS:
Overall Officials: Fathia Z. Zahran, PHD, Study Chair — Cairo University
Locations (1):
- Noha Nasr, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided